CLINICAL TRIAL: NCT00710021
Title: Effect of Vitamin D3 on the IFN Alpha Signature in Patients With Systemic Lupus Erythematosus (ALE02)
Brief Title: Vitamin D3 in Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ALE02
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Systemic Lupus Erythematosus; SLE; Lupus
Keywords: Systemic lupus erythematosus; SLE; Vitamin D3; Vitamin D deficiency; IFN alpha expression
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- vitamin D3 2000 IU (Experimental): Participants in this arm take a vitamin D3 dose of 2000 international units (IU) daily by mouth for a duration of 12 weeks.
  Interventions: Drug: Vitamin D3
- vitamin D3 4000 IU (Experimental): Participants in this arm take a vitamin D3 dose of 4000 international units (IU) daily by mouth for a duration of 12 weeks.
  Interventions: Drug: Vitamin D3
- vitamin D3 placebo (Placebo Comparator): Participants in this arm take a vitamin D3 placebo daily by mouth for a duration of 12 weeks.
  Interventions: Drug: Vitamin D3 placebo

INTERVENTIONS:
Drug: Vitamin D3 — 8% vitamin D3 powder, 84% microcrystalline cellulose, 8% fumed silica by weight
  Other Names: Cholecalciferol
  Arms: vitamin D3 2000 IU; vitamin D3 4000 IU
Drug: Vitamin D3 placebo — 86% microcrystalline cellulose, 14% fumed silica by weight
  Other Names: Cholecalciferol placebo
  Arms: vitamin D3 placebo

SUMMARY:
The purpose of this study is to explore the impact of vitamin D3 on the expression of alpha interferon (IFN alpha) expression in systemic lupus erythematosus (SLE) patients with vitamin D deficiency.

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is an autoimmune disease characterized by the production of autoantibodies with subsequent immune complex deposition and tissue inflammation. The role of interferon (IFN) alpha in the development of SLE has been repeatedly documented. Vitamin D deficiency is common among lupus patients. Vitamin D is recognized as a regulator of immune response. This study will explore the impact of vitamin D3 supplementation on IFN alpha expression in SLE patients.

The study will last approximately 12 weeks and consist of three treatment groups: 1.) Participants will receive vitamin D3 2000 IU daily 2.) Participants will receive vitamin D3 4000 IU daily 3.) Participants will receive a vitamin D3 placebo daily. There will be four study visits for each participant. Visits will occur at screening, study entry, and Weeks 6 and 12. Physical examination, vital signs, and blood and urine tests will occur at all visits. For females of childbearing potential, a pregnancy test will be performed at screening and Week 6.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE by American College of Rheumatology (ACR) criteria
* Serum 25-OH vitamin D level of 20 ng/mL or less
* Stable disease at screening, defined as a modified Safety of Estrogens in Lupus Erythematosus National Assessment SLE Disease Activity Index (SELENA-SLEDAI) of 4 or less
* Interferon (IFN) signature present. More information about this criterion can be found in the protocol
* Positive anti-double-stranded (anti-ds) DNA antibody blood test at screening
* If on corticosteroids, the dose must be less than 20 mg per day and stable for 4 weeks prior to screening and at study entry
* If on immunosuppressive or immunomodulatory medication such as azathioprine, methotrexate, leflunomide, mycophenolate, or hydroxychloroquine, the dose must be stable for 3 months prior to screening and at study entry
* If receiving a multivitamin or a vitamin D supplement, the dose of vitamin D must be 800 IU daily or less and stable for the 3 months prior to screening and at study entry
* Agree to use effective contraceptive methods for the duration of the study

Exclusion Criteria:

* Unwilling to stop using drugs or substances that may interfere with fat absorption
* Hypercalcemia
* Hypercalciuria
* History of hyperparathyroidism
* History of kidney stones
* History of cancer, except cervical carcinoma in situ and resected basal and squamous cell carcinomas of the skin
* Known history of chronic viral infections, including human immunodeficiency virus (HIV), Hepatitis B, and Hepatitis C
* Known active tuberculosis
* Any British Isles Lupus Assessment Group (BILAG) A or B manifestation with the exception of a BILAG B mucocutaneous manifestation
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) liver function tests greater than or equal to two times the upper limit of normal
* Dialysis or serum creatinine greater than 1.5 mg/dL
* Expectation by the investigator to increase corticosteroid or immunosuppressive or immunomodulatory medication dose at screening, study entry, or over the course of the study
* Treatment with cyclophosphamide within 3 months of screening
* Treatment with rituximab within 12 months of screening
* Other investigational drug and or treatment during the 4 weeks or seven half lives of the other investigational drug prior to study entry
* Drug or alcohol abuse within 6 months prior to study entry
* Treatment with digoxin
* Treatment with teriparatide
* Any condition that, in the opinion of the investigator, would jeopardize the subject's safety following exposure to the study drug
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Aranow, MD, Study Chair — Northwell Health; Diane Kamen, MD, Study Chair — Medical University of South Carolina
Locations (8):
- United States (8):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Feinstein Institute for Medical Research, Manhassett, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Data access is provided to the public in the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts that also provides data analysis tools available to researchers.

REFERENCES:
- [Background] Kamen DL, Cooper GS, Bouali H, Shaftman SR, Hollis BW, Gilkeson GS. Vitamin D deficiency in systemic lupus erythematosus. Autoimmun Rev. 2006 Feb;5(2):114-7. doi: 10.1016/j.autrev.2005.05.009. Epub 2005 Jun 21. PMID 16431339
- [Background] Mangini AJ, Lafyatis R, Van Seventer JM. Type I interferons inhibition of inflammatory T helper cell responses in systemic lupus erythematosus. Ann N Y Acad Sci. 2007 Jun;1108:11-23. doi: 10.1196/annals.1422.002. PMID 17893966
- [Background] Tan EM, Cohen AS, Fries JF, Masi AT, McShane DJ, Rothfield NF, Schaller JG, Talal N, Winchester RJ. The 1982 revised criteria for the classification of systemic lupus erythematosus. Arthritis Rheum. 1982 Nov;25(11):1271-7. doi: 10.1002/art.1780251101. PMID 7138600
- [Background] Hochberg MC. Updating the American College of Rheumatology revised criteria for the classification of systemic lupus erythematosus. Arthritis Rheum. 1997 Sep;40(9):1725. doi: 10.1002/art.1780400928. No abstract available. PMID 9324032
- [Background] Isenberg DA, Rahman A, Allen E, Farewell V, Akil M, Bruce IN, D'Cruz D, Griffiths B, Khamashta M, Maddison P, McHugh N, Snaith M, Teh LS, Yee CS, Zoma A, Gordon C. BILAG 2004. Development and initial validation of an updated version of the British Isles Lupus Assessment Group's disease activity index for patients with systemic lupus erythematosus. Rheumatology (Oxford). 2005 Jul;44(7):902-6. doi: 10.1093/rheumatology/keh624. Epub 2005 Apr 6. PMID 15814577
- [Result] Aranow C, Kamen DL, Dall'Era M, Massarotti EM, Mackay MC, Koumpouras F, Coca A, Chatham WW, Clowse ME, Criscione-Schreiber LG, Callahan S, Goldmuntz EA, Keyes-Elstein L, Oswald M, Gregersen PK, Diamond B. Randomized, Double-Blind, Placebo-Controlled Trial of the Effect of Vitamin D3 on the Interferon Signature in Patients With Systemic Lupus Erythematosus. Arthritis Rheumatol. 2015 Jul;67(7):1848-57. doi: 10.1002/art.39108. PMID 25777546
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: National Institute of Arthritis and Musculoskeletal and Skin Diseases: Handout on Health-System Lupus Erythematosus — https://www.niams.nih.gov/Health_Info/Lupus/default.asp
- Available data/document: Individual Participant Data Set: SDY474 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY474 — ImmPort study identifier is SDY474.
- Available data/document: Study Protocol: SDY474 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY474 — ImmPort study identifier is SDY474. The study protocol is located in the Design tab content.
- Available data/document: Study summary, -design, -adverse event(s), -meds,-demographics, -lab tests, -mechanistic assays, - files: SDY474 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY474 — ImmPort study identifier is SDY474.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received a 12-week course of oral vitamin D3-placebo (cholecalciferol placebo, 1 dose daily).
- Vitamin D3 2000 IU: Participants received a 12-week course of oral Vitamin D3 (cholecalciferol, 2,000 international units [IU] daily).
- Vitamin D3 4000 IU: Participants received a 12-week course of oral vitamin D3 (cholecalciferol, 4,000 IU daily).
Period: Overall Study
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU
Started | 19 | 19 | 19
Modified Intent-to-Treat (mITT) | 19 | 17 (2 subjects who did not take study drug were excluded from mITT) | 18 (1 subject who did not take study drug was excluded from mITT)
Completed | 18 | 16 | 18
Not Completed | 1 | 3 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Subject's Decision | 0 | 1 | 0
Not completed — Subject misrandomized | 0 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Total
Number analyzed (Participants) | 19 | 17 | 18 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (12.3) | 36.5 (10.9) | 38.3 (12.9) | 37.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 16 | 51
  Male | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 19 | 17 | 18 | 54
Years with Systemic Lupus Erythematosus (SLE) at Baseline [Mean (Standard Deviation); unit: years] — Years since systemic lupus erythematosus was diagnosed by a physician. This information was obtained by medical history during the Baseline visit.
  years | 10.9 (7.8) | 10.0 (7.8) | 8.7 (6.0) | 9.9 (7.1)
Number of American College of Rheumatology (ACR) Criteria met at Screening [Mean (Standard Deviation); unit: number of criteria met] — The diagnosis of SLE is made using the American College of Rheumatology (ACR) criteria. The presence of 4 or more of the following 11 ACR criteria is diagnostic for lupus and was required to participate in this trial: malar rash, discoid rash, photosensitive skin rash, oral ulcers, nonerosive arthritis, pleuritis/pericarditis, renal disorder, neurologic disorder, hematologic disorder, immunologic disorder, and a positive antinuclear antibody (ANA) test. Reference: Arthritis Rheum 1997; 40(9): 1725.
  number of criteria met | 5.4 (1.3) | 5.5 (1.1) | 5.8 (1.3) | 5.6 (1.2)
Modified SELENA-SLEDAI Score [Mean (Standard Deviation); unit: score] — The modified Safety of Estrogens in Lupus Erythematosus National Assessment SLE Disease Activity Index (SELENA-SLEDAI) is calculated from 24 individual descriptors; scores may range from 0 (indicates inactive disease) to 105 (the maximum theoretical score). The SELENA-SLEDAI assesses disease activity for 10 days prior to and including the day of assessment. For this study, the SELENA-SLEDAI score was modified to include proteinuria defined by dipstick rather than 24 hour urine. A SELENA-SLEDAI score of 4 or less, indicative of stable disease, was a requirement to enter this study.
  score | 2.9 (1.2) | 2.7 (1.2) | 2.6 (1.0) | 2.7 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With an IFN Alpha Signature Response at Week 12
Description: Presence of an Interferon (IFN) Alpha signature response is defined as: a reduction in expression from baseline (Screening) of at least 50% for 1 of 3 IFN Alpha responsive genes (Ifit1, Ifi44, Mx1) with concurrent expression in the remaining 2 genes at a level not more than 25% above baseline, or a reduction in expression from baseline of at least 25% for 2 of the 3 IFN Alpha responsive genes with concurrent expression in the third gene at a level of no more than 25% above baseline. Gene expression was measured on peripheral blood samples using qRT-PCR. Missing data were considered as response failures during calculation.
Time Frame: 0, Week 12
Population: Modified Intent-to-Treat. Although presence of a positive IFN Alpha Signature at the Screening visit was an entry criterion for the study, 8 subjects (4 Placebo, 2 Vitamin D3 2000 IU, 2 Vitamin D3 4000 IU ) who did not have a signature were included in the study.
Measure: Number; unit: Percent of participants
Groups:
- Vitamin D3 2000 and 4000 IU (Pooled ): This is a statistically pooled group of those participants randomized to either vitamin D3 2,000 IU or vitamin D3 4,000 IU treatment (e.g., pooled group for statistical analysis purposes only).
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 19 | 17 | 18 | 35
Percent of participants | 36.8 | 23.5 | 27.8 | 25.7
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.53, Fisher Exact — The p-value compares the Placebo with the pooled Vitamin D treatment group

2. Secondary Outcome: Percent of Participants With an IFN Alpha Signature Response at Week 6
Description: as for outcome 1
Time Frame: 0, Week 6
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 19 | 17 | 18 | 35
Percent of participants | 36.8 | 17.6 | 5.6 | 11.4
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.038, Fisher Exact — The p-value compares the Placebo with the pooled Vitamin D treatment group

3. Secondary Outcome: Percent of Participants With IFN Alpha Signature at Week 12
Description: An Interferon (IFN) Alpha signature is defined as: expression of Mx1, Ifit1, or Ifi44 at a level greater than or equal to 4 standard deviations above the mean of a set of normal controls, or expression of 2 of the 3 genes at a level greater than or equal to 2 standard deviations above the mean of a set of normal controls. Gene expression was measured on peripheral blood samples using qRT-PCR. Missing data were assumed as signatures during calculation.
Time Frame: 0, Week 12
Population: Modified Intent-to-Treat. Although presence of a positive IFN Alpha Signature at the Screening visit was an entry criterion for the study, 8 subjects (4 Placebo, 2 Vitamin D3 2000 IU, 2 Vitamin D3 4000 IU) who did not have a signature were included in the study.
Measure: Number; unit: Percent of participants
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 19 | 17 | 18 | 35
Percent of participants | 78.9 | 94.1 | 100.0 | 97.1
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.047, Fisher Exact — The p-value compares the Placebo with the pooled Vitamin D treatment group

4. Secondary Outcome: Percent of Participants With IFN Alpha Signature at Week 6
Description: as for outcome 3
Time Frame: Week 6
Population: as for outcome 3
Measure: Number; unit: Percent of participants
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 19 | 17 | 18 | 35
Percent of participants | 84.2 | 94.1 | 100.0 | 97.1
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.12, Fisher Exact — The p-value compares the Placebo with the pooled Vitamin D treatment group

5. Secondary Outcome: qRT-PCR Fold Change in Ifit1 Gene Expression From Baseline to Week 12
Description: The Ifit1 gene is one of three genes included in the definition of the alpha-interferon signature used for this study. This gene encodes an interferon-induced protein with tetratricopeptide repeats. Quantitative real-time polymerase chain reaction (qRT-PCR) was used to measure gene expression in peripheral blood mononuclear cells obtained by blood draw. Gene expression is quantified as "fold change" relative to normal controls and is computed using a comparative CT (threshold cycle) method. A study hypothesis was that expression of alpha-interferon signature genes would decrease with increasing vitamin D levels. A decrease in gene expression from baseline to Week 12 is represented as a negative value (and vice versa).
Time Frame: 0, Week 12
Population: Modified Intent-to-Treat with available data
Measure: Mean (Standard Deviation); unit: qRT-PCR fold change
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 15 | 15 | 18 | 33
qRT-PCR fold change | -8.6 (40.5) | -2.9 (57.0) | 5.2 (33.9) | 1.5 (45.3)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.31, F-tests derived from the GLM — The p-value compares the Placebo with the pooled Vitamin D treatment group; The test was for the comparison of pooled Vitamin D versus Placebo after adjustment for baseline Ifit1 expression

6. Secondary Outcome: qRT-PCR Fold Change in Ifit1 Gene Expression From Baseline to Week 6
Description: The Ifit1 gene is one of three genes included in the definition of the alpha-interferon signature used for this study. It encodes an interferon-induced protein with tetratricopeptide repeats. Quantitative real-time polymerase chain reaction (qRT-PCR) was used to measure gene expression in peripheral blood mononuclear cells obtained by blood draw. Gene expression is quantified as "fold change" relative to normal controls and is computed using a comparative CT (threshold cycle) method. A study hypothesis was that expression of alpha-interferon signature genes would decrease with increasing vitamin D levels. A decrease in gene expression from baseline to Week 6 is represented as a negative value (and vice versa).
Time Frame: 0, Week 6
Population: Modified Intent-to-Treat with available data
Measure: Mean (Standard Deviation); unit: qRT-PCR fold change
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 16 | 13 | 17 | 30
qRT-PCR fold change | -15.5 (38.0) | -11.6 (35.5) | 6.3 (18.1) | -1.4 (28.0)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.019, F-tests derived from the GLM — The p-value compares the Placebo with the pooled Vitamin D treatment group; The test was for the comparison of pooled Vitamin D versus Placebo after adjustment for baseline Ifit1 expression

7. Secondary Outcome: qRT-PCR Fold Change in Ifi44 Gene Expression From Baseline to Week 12
Description: The Ifi44 gene is one of three genes included in the definition of the alpha-interferon signature used for this study. It encodes interferon-induced protein 44. Quantitative real-time polymerase chain reaction (qRT-PCR) was used to measure gene expression in peripheral blood mononuclear cells obtained by blood draw. Gene expression is quantified as "fold change" relative to normal controls and is computed using a comparative CT (threshold cycle) method. A study hypothesis was that expression of alpha-interferon signature genes would decrease with increasing vitamin D levels. A decrease in gene expression from baseline to Week 12 is represented as a negative value (and vice versa).
Time Frame: 0, Week 12
Population: Modified Intent-to-Treat with available data
Measure: Mean (Standard Deviation); unit: qRT-PCR fold change
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 15 | 15 | 18 | 33
qRT-PCR fold change | -2.5 (16.4) | -0.3 (9.8) | 2.9 (11.7) | 1.4 (10.8)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.28, F-tests derived from the GLM — The p-value compares the Placebo with the pooled Vitamin D treatment group; The test was for the comparison of pooled Vitamin D versus Placebo after adjustment for baseline Ifi44 expression

8. Secondary Outcome: qRT-PCR Fold Change in Ifi44 Gene Expression From Baseline to Week 6
Description: The Ifi44 gene is one of three genes included in the definition of the alpha-interferon signature used for this study. It encodes interferon-induced protein 44. Quantitative real-time polymerase chain reaction (qRT-PCR) was used to measure gene expression in peripheral blood mononuclear cells obtained by blood draw. Gene expression is quantified as "fold change" relative to normal controls and is computed using a comparative CT (threshold cycle) method. A study hypothesis was that expression of alpha-interferon signature genes would decrease with increasing vitamin D levels. A decrease in gene expression from baseline to Week 6 is represented as a negative value (and vice versa).
Time Frame: 0, Week 6
Population: Modified Intent-to-Treat with available data
Measure: Mean (Standard Deviation); unit: qRT-PCR fold change
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 16 | 13 | 17 | 30
qRT-PCR fold change | -3.9 (12.8) | -4.6 (11.0) | 4.1 (5.9) | 0.3 (9.4)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.050, F-tests derived from the GLM — The p-value compares the Placebo with the pooled Vitamin D treatment group; The test was for the comparison of pooled Vitamin D versus Placebo after adjustment for baseline Ifi44 expression

9. Secondary Outcome: qRT-PCR Fold Change in Mx1 Gene Expression From Baseline to Week 12
Description: The Mx1 gene is one of three genes included in the definition of the alpha-interferon signature used for this study. It encodes for the homolog of mouse myxovirus (influenza virus) resistance 1 protein. Quantitative real-time polymerase chain reaction (qRT-PCR) was used to measure gene expression in peripheral blood mononuclear cells obtained by blood draw. Gene expression is quantified as "fold change" relative to normal controls and is computed using a comparative CT (threshold cycle) method. A study hypothesis was that expression of alpha-interferon signature genes would decrease with increasing vitamin D levels. A decrease in gene expression from baseline to Week 12 is represented as a negative value (and vice versa).
Time Frame: 0, Week 12
Population: Modified Intent-to-Treat with available data
Measure: Mean (Standard Deviation); unit: qRT-PCR fold change
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 15 | 15 | 18 | 33
qRT-PCR fold change | -1.6 (14.0) | 2.0 (12.5) | 4.8 (11.6) | 3.5 (11.9)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.29, F-tests derived from the GLM — The p-value compares the Placebo with the pooled Vitamin D treatment group; The test was for the comparison of pooled Vitamin D versus Placebo after adjustment for baseline Mx1 expression

10. Secondary Outcome: qRT-PCR Fold Change in Mx1 Gene Expression From Baseline to Week 6
Description: The Mx1 gene is one of three genes included in the definition of the alpha-interferon signature used for this study. It encodes for the homolog of mouse myxovirus (influenza virus) resistance 1 protein. Quantitative real-time polymerase chain reaction (qRT-PCR) was used to measure gene expression in peripheral blood mononuclear cells obtained by blood draw. Gene expression is quantified as "fold change" relative to normal controls and is computed using a comparative CT (threshold cycle) method. A study hypothesis was that expression of alpha-interferon signature genes would decrease with increasing vitamin D levels. A decrease in gene expression from baseline to Week 6 is represented as a negative value (and vice versa).
Time Frame: 0, Week 6
Population: Modified Intent-to-Treat with available data
Measure: Mean (Standard Deviation); unit: qRT-PCR fold change
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 16 | 13 | 17 | 30
qRT-PCR fold change | -4.8 (10.5) | 1.4 (19.5) | 0.7 (6.7) | 1.0 (13.5)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.014, F-tests derived from the GLM — The p-value compares the Placebo with the pooled Vitamin D treatment group; The test was for the comparison of pooled Vitamin D versus Placebo after adjustment for baseline Mx1 expression

11. Secondary Outcome: Change in Serum C3 Level From Baseline to Week 12
Description: C3 is a blood test that measures the activity of the complement component 3 (C3) protein. The normal C3 range is 75 to 135 mg/dL. Patients with active systemic lupus erythematosus may have a lower-than-normal level of C3. A decrease in C3 level over time may indicate disease activity. An increase in C3 from baseline to Week 12 is represented as a positive value (and vice versa).
Time Frame: 0, Week 12
Population: Modified Intent-to-Treat with available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 18 | 16 | 18 | 34
mg/dL | 1.8 (16.1) | 0.7 (11.1) | 2.9 (11.1) | 1.9 (11.0)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.96, F-tests derived from the GLM — The p-value compares the Placebo with the pooled Vitamin D treatment group; The test was for the comparison of pooled Vitamin D versus Placebo after adjustment for baseline serum C3 level

12. Secondary Outcome: Change in Serum C3 Level From Baseline to Week 6
Description: C3 is a blood test that measures the activity of the complement component 3 (C3) protein. The normal C3 range is 75 to 135 mg/dL. Patients with active systemic lupus erythematosus may have a lower-than-normal level of C3. A decrease in C3 level over time may indicate disease activity. An increase in C3 from baseline to Week 6 is represented as a positive value (and vice versa).
Time Frame: 0, Week 6
Population: Modified Intent-to-Treat with available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 19 | 15 | 18 | 33
mg/dL | 3.3 (10.9) | 3.8 (11.2) | 3.7 (10.3) | 3.8 (10.5)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.67, F-tests derived from the GLM — The p-value compares the Placebo with the pooled Vitamin D treatment group; The test was for the comparison of pooled Vitamin D versus Placebo after adjustment for baseline serum C3 level

13. Secondary Outcome: Change in Serum C4 Level From Baseline to Week 12
Description: C4 is a blood test that measures the activity of the complement component 4 (C4) protein. The normal range for males is 12 to 72 mg/dL and the normal range for females is 13 to 75 mg/dL. Patients with active systemic lupus erythematosus may have a lower-than-normal level of C4. A decrease in C4 level over time may indicate disease activity. An increase in C4 from baseline to Week 12 is represented as a positive value (and vice versa).
Time Frame: 0, Week 12
Population: Modified Intent-to-Treat with available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 18 | 16 | 18 | 34
mg/dL | 0.2 (2.5) | -0.3 (2.9) | 1.9 (4.4) | .9 (3.9)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.59, F-tests derived from the GLM — The p-value compares the Placebo with the pooled Vitamin D treatment group; The test was for the comparison of pooled Vitamin D versus Placebo after adjustment for baseline serum C4 level

14. Secondary Outcome: Change in Serum C4 Level From Baseline to Week 6
Description: Outcome measure description: C4 is a blood test that measures the activity of the complement component 4 (C4) protein. The normal range for males is 12 to 72 mg/dL and the normal range for females is 13 to 75 mg/dL. Patients with active systemic lupus erythematosus may have a lower-than-normal level of C4. A decrease in C4 level over time may indicate disease activity. An increase in C4 from baseline to Week 6 is represented as a positive value (and vice versa).
Time Frame: 0, Week 6
Population: Modified Intent-to-Treat with available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 19 | 15 | 18 | 33
mg/dL | 0.3 (3.3) | -0.8 (2.7) | 0.4 (2.8) | -0.2 (2.7)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.65, F-tests derived from the GLM — The p-value compares the Placebo with the pooled Vitamin D treatment group; The test was for the comparison of pooled Vitamin D versus Placebo after adjustment for baseline serum C4 level

15. Secondary Outcome: Change in Status for Anti-double-stranded DNA Autoantibody From Baseline to Week 12
Description: Patients with systemic lupus erythematosus (SLE) may have autoantibodies (e.g., self against self) to double-stranded DNA. Double-stranded DNA is one of multiple diagnostic tests for SLE and levels may be associated with disease activity. A positive test for autoantibodies to double-stranded DNA is based on the normal range from the local laboratory. Change in status (+ or -) from baseline is evaluated.
Time Frame: 0, Week 12
Population: Modified Intent-to-Treat with available data
Measure: Number; unit: Percent of participants
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 17 | 16 | 18 | 34
Percent of participants
  Positive at Baseline, Positive at Week 12 | 94.1 | 100.0 | 77.8 | 88.2
  Positive at Baseline, Negative at Week 12 | 0.0 | 0.0 | 11.0 | 6.0
  Negative at Baseline, Positive at Week 12 | 0.0 | 0.0 | 5.6 | 2.9
  Negative at Baseline, Negative at Week 12 | 5.9 | 0.0 | 5.6 | 2.9
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.86, Fisher Exact — The p-value compares the Placebo with the pooled Vitamin D treatment group

16. Secondary Outcome: Change in Status for Anti-double-stranded DNA Autoantibody From Baseline to Week 6
Description: as for outcome 15
Time Frame: 0, Week 6
Population: Modified Intent-to-Treat with available data
Measure: Number; unit: Percent of participants
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 19 | 16 | 18 | 34
Percent of participants
  Positive at Baseline, Positive at Week 6 | 94.7 | 93.7 | 88.9 | 91.2
  Positive at Baseline, Negative at Week 6 | 0.0 | 6.3 | 0.0 | 2.9
  Negative at Baseline, Positive at Week 6 | 0.0 | 0.0 | 0.0 | 0.0
  Negative at Baseline, Negative at Week 6 | 5.3 | 0.0 | 11.1 | 5.9
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 1.0, Fisher Exact — The p-value compares the Placebo with the pooled Vitamin D treatment group

17. Secondary Outcome: Change in SELENA-SLEDAI Total Score From Baseline to Week 12
Description: The modified Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus (SLE) Disease Activity Index (SELENA-SLEDAI) score is a weighted scale score ranging from 0 to 105 based on the presence or absence of 24 manifestations of SLE. The SELENA-SLEDAI assesses disease activity for 10 days prior to and including the day of assessment. For this study, the SELENA-SLEDAI score was modified to include proteinuria defined by dipstick rather than 24 hour urine. Positive change in the SELENA-SLEDAI score indicate increased disease activity.
Time Frame: 0, Week 12
Population: Modified Intent-to-Treat with available data
Measure: Mean (Standard Deviation); unit: Change in Scores on a Scale
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 18 | 16 | 18 | 34
Change in Scores on a Scale | 0.0 (0.7) | 0.2 (1.8) | 0.2 (1.9) | 0.2 (1.8)
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.62, F-tests derived from the GLM — The p-value compares the Placebo with the pooled Vitamin D treatment group; The test was for the comparison of pooled Vitamin D versus Placebo after adjustment for baseline SELENA-SLEDAI score

18. Secondary Outcome: Cardiorespiratory BILAG Status at Week 12
Description: The British Isles Lupus Assessment Group (BILAG) assessment gives a grade for each of 9 body systems (e.g., domains). Grades reflect systemic lupus erythematosus disease activity as follows: A (severe), B (moderate), C (mild), D (inactive at present but previously affected), E (inactive and system never involved). To be randomized, subjects had to have mild or inactive disease (C,D,E) in all but the mucocutaneous system in which B(moderate) disease was also allowed. The percent of subjects experiencing A or B level activity at Week 12 is assessed for the "Cardiorespiratory-specific" body system.
Time Frame: Week 12
Population: Modified Intent-to-Treat with available data
Measure: Number; unit: Percent with grade A or B
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 18 | 16 | 18 | 34
Percent with grade A or B | 0.0 | 6.3 | 0.0 | 2.9
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 1.0, Fisher Exact — The p-value compares the Placebo with the pooled Vitamin D treatment group

19. Secondary Outcome: Constitutional BILAG Status at Week 12
Description: The British Isles Lupus Assessment Group (BILAG) assessment gives a grade for each of 9 body systems (e.g., domains). Grades reflect systemic lupus erythematosus disease activity as follows: A (severe), B (moderate), C (mild), D (inactive at present but previously affected), E (inactive and system never involved). To be randomized, subjects had to have mild or inactive disease (C,D,E) in all but the mucocutaneous system in which B(moderate) disease was also allowed. The percent of subjects experiencing A or B level activity at Week 12 is assessed for the "Constitutional-specific" body system.
Time Frame: Week 12
Population: Modified Intent-to-Treat with available data
Measure: Number; unit: Percent with grade A or B
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 18 | 16 | 18 | 34
Percent with grade A or B | 0.0 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 1.0, Fisher Exact — The p-value compares the Placebo with the pooled Vitamin D treatment group

20. Secondary Outcome: Gastrointestinal BILAG Status at Week 12
Description: The British Isles Lupus Assessment Group (BILAG) assessment gives a grade for each of 9 body systems (e.g., domains). Grades reflect systemic lupus erythematosus disease activity as follows: A (severe), B (moderate), C (mild), D (inactive at present but previously affected), E (inactive and system never involved). To be randomized, subjects had to have mild or inactive disease (C,D,E) in all but the mucocutaneous system in which B(moderate) disease was also allowed. The percent of subjects experiencing A or B level activity at Week 12 is assessed for the "Gastrointestinal-specific" body system.
Time Frame: Week 12
Population: Modified Intent-to-Treat with available data
Measure: Number; unit: Percent with grade A or B
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 18 | 16 | 18 | 34
Percent with grade A or B | 0.0 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 1.0, Fisher Exact — The p-value compares the Placebo with the pooled Vitamin D treatment group

21. Secondary Outcome: Hematological BILAG Status at Week 12
Description: The British Isles Lupus Assessment Group (BILAG) assessment gives a grade for each of 9 body systems (e.g., domains). Grades reflect systemic lupus erythematosus disease activity as follows: A (severe), B (moderate), C (mild), D (inactive at present but previously affected), E (inactive and system never involved). To be randomized, subjects had to have mild or inactive disease (C,D,E) in all but the mucocutaneous system in which B(moderate) disease was also allowed. The percent of subjects experiencing A or B level activity at Week 12 is assessed for the "Hematological-specific" body system.
Time Frame: Week 12
Population: Modified Intent-to-Treat with available data
Measure: Number; unit: Percent with grade A or B
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 18 | 16 | 18 | 34
Percent with grade A or B | 0.0 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 1.0, Fisher Exact — The p-value compares the Placebo with the pooled Vitamin D treatment group

22. Secondary Outcome: Mucocutaneous BILAG Status at Week 12
Description: The British Isles Lupus Assessment Group (BILAG) assessment gives a grade for each of 9 body systems (e.g., domains). Grades reflect systemic lupus erythematosus disease activity as follows: A (severe), B (moderate), C (mild), D (inactive at present but previously affected), E (inactive and system never involved). To be randomized, subjects had to have mild or inactive disease (C,D,E) in all but the mucocutaneous system in which B(moderate) disease was also allowed. The percent of subjects experiencing A or B level activity at Week 12 is assessed for the "Mucocutaneous-specific" body system.
Time Frame: Week 12
Population: Modified Intent-to-Treat with available data
Measure: Number; unit: Percent with grade A or B
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 18 | 16 | 18 | 34
Percent with grade A or B | 5.6 | 12.5 | 0.0 | 5.9
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 1.0, Fisher Exact — The p-value compares the Placebo with the pooled Vitamin D treatment group

23. Secondary Outcome: Musculoskeletal BILAG Status at Week 12
Description: Outcome measure description: The British Isles Lupus Assessment Group (BILAG) assessment gives a grade for each of 9 body systems (e.g., domains). Grades reflect systemic lupus erythematosus disease activity as follows: A (severe), B (moderate), C (mild), D (inactive at present but previously affected), E (inactive and system never involved). To be randomized, subjects had to have mild or inactive disease (C,D,E) in all but the mucocutaneous system in which B(moderate) disease was also allowed. The percent of subjects experiencing A or B level activity at Week 12 is assessed for the "Musculoskeletal-specific" body system.
Time Frame: Week 12
Population: Modified Intent-to-Treat with available data
Measure: Number; unit: Percent with grade A or B
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 18 | 16 | 18 | 34
Percent with grade A or B | 5.6 | 0.0 | 11.1 | 5.9
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 1.0, Fisher Exact — The p-value compares the Placebo with the pooled Vitamin D treatment group

24. Secondary Outcome: Neuropsychiatric BILAG Status at Week 12
Description: The British Isles Lupus Assessment Group (BILAG) assessment gives a grade for each of 9 body systems (e.g., domains). Grades reflect systemic lupus erythematosus disease activity as follows: A (severe), B (moderate), C (mild), D (inactive at present but previously affected), E (inactive and system never involved). To be randomized, subjects had to have mild or inactive disease (C,D,E) in all but the mucocutaneous system in which B(moderate) disease was also allowed. The percent of subjects experiencing A or B level activity at Week 12 is assessed for the "Neuropsychiatric-specific" body system.
Time Frame: Week 12
Population: Modified Intent-to-Treat with available data
Measure: Number; unit: Percent with grade A or B
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 18 | 16 | 18 | 34
Percent with grade A or B | 0.0 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 1.0, Fisher Exact — The p-value compares the Placebo with the pooled Vitamin D treatment group

25. Secondary Outcome: Ophthalmic BILAG Status at Week 12
Description: The British Isles Lupus Assessment Group (BILAG) assessment gives a grade for each of 9 body systems (e.g., domains). Grades reflect systemic lupus erythematosus disease activity as follows: A (severe), B (moderate), C (mild), D (inactive at present but previously affected), E (inactive and system never involved). To be randomized, subjects had to have mild or inactive disease (C,D,E) in all but the mucocutaneous system in which B(moderate) disease was also allowed. The percent of subjects experiencing A or B level activity at Week 12 is assessed for the "Ophthalmic-specific" body system.
Time Frame: Week 12
Population: Modified Intent-to-Treat with available data
Measure: Number; unit: Percent with grade A or B
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 18 | 16 | 18 | 34
Percent with grade A or B | 0.0 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 1.0, Fisher Exact — The p-value compares the Placebo with the pooled Vitamin D treatment group

26. Secondary Outcome: Renal BILAG Status at Week 12
Description: The British Isles Lupus Assessment Group (BILAG) assessment gives a grade for each of 9 body systems (e.g., domains). Grades reflect systemic lupus erythematosus disease activity as follows: A (severe), B (moderate), C (mild), D (inactive at present but previously affected), E (inactive and system never involved). To be randomized, subjects had to have mild or inactive disease (C,D,E) in all but the mucocutaneous system in which B(moderate) disease was also allowed. The percent of subjects experiencing A or B level activity at Week 12 is assessed for the "Renal-specific" body system.
Time Frame: Week 12
Population: Modified Intent-to-Treat with available data
Measure: Number; unit: Percent with grade A or B
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 18 | 16 | 18 | 34
Percent with grade A or B | 0.0 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 1.0, Fisher Exact — The p-value compares the Placebo with the pooled Vitamin D treatment group

27. Secondary Outcome: Percent of Participants With Adverse Events of Grade 3 or Above
Description: Grades are based on National Cancer Institute--Common Terminology Criteria (NCI-CTCAE) Version 3.0 over the duration of the study. Participants who experienced at least one grade 3 or higher adverse event (AE) are counted only once. The adverse events are treatment-emergent, which means that the AE occurred after taking the first dose of study drug.
Time Frame: From start of study treatment through Week 12
Population: Safety
Measure: Number; unit: Percent of participants
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU | Vitamin D3 2000 and 4000 IU (Pooled )
Number analyzed (Participants) | 19 | 17 | 18 | 35
Percent of participants | 5.3 | 23.5 | 22.2 | 22.9
Statistical Analysis 1: Comparison: Placebo vs Vitamin D3 2000 and 4000 IU (Pooled ); Test type: Superiority or Other; p = 0.10, Cochran-Mantel-Haenszel — The p-value compares the Placebo with the pooled Vitamin D treatment group; Note that none of the Grade 3 or above events were considered by the investigators to be related to study treatment

ADVERSE EVENTS:
Time Frame: Baseline to 12 weeks
Description: This study graded the severity of adverse events experienced by the study participant according to criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.0 (June 10, 2003)
Arm/Group | Placebo | Vitamin D3 2000 IU | Vitamin D3 4000 IU
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17 | 3/18
Other Adverse Events (participants affected / at risk) | 15/19 | 16/17 | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Vitamin D3 2000 IU (N=17) | Vitamin D3 4000 IU (N=18)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Vitamin D3 2000 IU (N=17) | Vitamin D3 4000 IU (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Blood albumin decreased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Blood glucose decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 4 (4) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 4 (4) | 3 (3) | 5 (5)
Lymphocyte count decreased (Investigations) | 3 (3) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 3 (3) | 5 (5)
White blood cell count decreased (Investigations) | 6 (7) | 2 (2) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No